CLINICAL TRIAL: NCT05945251
Title: Individualized Online Cognitive Behavioral Therapy for Children With Functional Abdominal Pain Disorders - the Child's Pain Regulation
Brief Title: ICBT for Children With FAPDs - the Child's Pain Regulation
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Child and Adolescent Psychiatry, Stockholm (Industry)
Responsible Party: Principal Investigator, Maria Lalouni, Assistant Professor, Karolinska Institutet
Other Study IDs: 20223238
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Functional Abdominal Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FAPDs: Children 8-17 years with FAPDs
  Interventions: Other: Internet-delivered cognitive behavioral therapy
- Controls: Children 8-17 years without FAPDs

INTERVENTIONS:
Other: Internet-delivered cognitive behavioral therapy — Ten weekly modules for children and ten weekly modules for parents. Exposure-based cognitive behavioral therapy delivered online with asynchronous support via text messages from psychologists.
  Groups: FAPDs

SUMMARY:
Functional abdominal pain disorders (FAPDs) in children are common (14%) and abdominal pain has increased rapidly in children during the last ten years in Sweden. Many children with FAPDs have low quality of life, missed school days, and about 30-40% suffer from psychiatric comorbidity. FAPDs are often sustained into adulthood and a large Swedish cohort study showed that abdominal pain during childhood is an independent strong predictor anxiety and depression later in life. Internet-cognitive behavioral therapy (Internet-CBT) can improve FAPD symptoms, but a significant number of children does not respond to the treatment.

We will here determine the pain regulation in children with FAPDs, compared with healthy controls, and assess:

What aspects of the child's pain regulation is related to improvement for children with FAPDs engaging in Internet-CBT?

Does some aspects of the child's pain regulation change during treatment?

ELIGIBILITY:
Inclusion Criteria:

Children 8-17 years with FAPDs: Have been offered treatment at BUP Internetbehandling for FAPDs.

Children 8-17 years without FAPDs: Not affected by recurrent (every week) or persistant pain during the last year.

Exclusion Criteria:

Contraindication for MR (metal implant or metal object in body, claustrophobia, pregnancy)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children (n=40) aged 8-17 with FAPDs who are patients at BUP Internetbehandling within the Child and Adolescent Psychiatry in Stockholm will be included in the study. Their behavioral and neural pain mechanisms will be assessed before and after Internet-CBT. We will also recruit healthy control children (n=40) aged 8-17 to compare the pain regulation between the groups. First, we will ask whether there are healthy siblings to the participating children with FAPDs that are willing to participate. If we don't get enough children by asking siblings, social media will be used in the recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold on navel | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Algometer pressure (in kPa) for the pain threshold
Unpleasantness of pressure pain threshold on navel | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Children rate their unpleasantness on a scale 0-10

SECONDARY OUTCOMES:
Pressure pain threshold on thigh | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Algometer pressure (in kPa) for the pain threshold
Unpleasantness of pressure pain threshold on thigh | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Children rate their unpleasantness on a scale 0-10
Conditioned pain modulation | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Conditioned pain: hand in 10°C cold water, test pain: presseure pain thresholds by algometer on the participant's thigh. Difference in pressure pain thresholds with and without the simultaneous conditioned stimuli
Temporal summation | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Pinprick stimuli of low pain, one time, then repeated 10 times. Pain after repeated stimulus minus pain for the single stimulus.
Sensory attenuation of pain | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Pressure pain thresholds (kPa) applied by the child or the experimenter. Sensory attenuation = difference in pain threshold between self-induced and experimenter induced
Resting state fMRI | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Differences in network connectivity (Yeo networks + subcortical areas) and between seed (trunk in the somatosensory cortex) to Yeo brain networks + subcortical areas).
fMRI during low pain compared with non-painful tactile stimulus | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Differences in network connectivity (Yeo networks + subcortical areas) and between seed (trunk in the somatosensory cortex) to Yeo brain networks + subcortical areas).
Pediatric Quality of Life Inventory Gastrointestinal Symptom Scale (PedsQL Gastro) | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Self-assessed questionnaire of abdominal symptoms
Faces Pain Rating Scale (FACES) | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Self-assessed questionnaire of pain intensity
Visceral sensitivity Index, child-adapted short version (VSI-C) | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Self-assessed questionnaire of gastrointestinal-specific anxiety
Irritable bowel syndrome-behavioral responses questionnaire, child-adapted short version (BRQ-C) | Baseline differences and baseline to follow-up after 10 week's treatment (or 10 week's wait for healthy children)
  Self-assessed questionnaire of gastrointestinal-specific avoidance and controlling behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lalouni, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Karolinska Institutet, Sweden